CLINICAL TRIAL: NCT07166653
Title: Nordic Digital Health Education as an Implementation Tool for Hospital-at-home - Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Hospital-at-Home Education as Implementation Tool - RCT
Acronym: HAH-EDUCATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Lund University (Other); University College Copenhagen (Other); Ostfold University College (Other); Region Capital Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NorDigHE HaH RCT Protocol
Record Dates: First submitted 2025-08-08; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Hospital
Keywords: clinical competence; digital health; education; hospital at home; hospital in the home; implementation; telemedicine

STUDY DESIGN:
Intervention Model Description: The study is designed as a two-armed, multicenter, superiority, cluster-randomized clinical trial with the hospital as the unit of randomization. The participating hospitals will autonomously select the relevant clinical departments and related staff to undergo the education tested. Data are collected at baseline, after 3, and 6 months. The intervention group also collects a 12-month maintenance assessment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group receives the NorDigHE HaH education embedded in the WHO Fast-IM.
  Interventions: Behavioral: HaH education
- Control group (No Intervention): The control group continues treatment as usual over a 6-month period. To enhance participant retention, the control group will be offered the education after study completion and as a quality initiative.

INTERVENTIONS:
Behavioral: HaH education — The intervention consists of the online NorDigHE HaH education with tailored implementation tools em-bedded in the WHO Fast-IM. The education is delivered online and asynchronously, combining e-learning, simulations, reflection exercises, and practical task training.
  The trial has adopted the evidence-based WHO Fast-track Implementation Model (WHO Fast-IM) as a framework to support the effectiveness and reporting of the implementation, and the tailored implementation tools embedded in the model will be provided as part of the intervention to support in-tegration into daily clinical routines. The tailored toolbox consists of workshops, introductory meetings, written guides, and access to a hotline staffed by project specialists to facilitate implementation.
  Other Names: NorDigHE education
  Arms: Intervention group

SUMMARY:
To enhance implementation of Hospital-at-home (HaH) in Scandinavia, the Nordic Digital Health & Education (NorDigHE) project has developed a comprehensive virtual education on HaH for clinical staff. The goal of this clinical trial is to evaluate whether an online education for clinical staff can enhance the implementation of HaH services in hospitals across Denmark, Norway, and Sweden.

The primary outcome of the RCT is HaH implementation measured at organization level, understood as a change in clinical practice by increased HaH activity. Secondary outcomes are HaH knowledge and motivation among clinical staff as well as patient days in hospital, days hospitalized at home, 30-day readmission, and mortality.

Researchers will compare hospitals receiving the NorDigHE education (intervention group) to hospitals continuing treatment as usual (control group) to see if the education leads to greater adoption of HaH and changes in service delivery.

Participants will:

* Complete baseline, 3-month, and 6-month surveys assessing HaH activity, staff knowledge, and motivation.
* Participate in a 12-month follow-up assessment (intervention group only).
* Be invited (patients, staff, and management) to take part in semi-structured interviews to share experiences and preferences related to HaH.
* (For staff in the intervention group) Complete the NorDigHE virtual education program embedded in the WHO Fast-IM.

After the study, the control group will be offered access to the NorDigHE education as a participant retention measure.

DETAILED DESCRIPTION:
Background: In response to increasing pressures on healthcare systems due to aging populations, and increasing shortages of clinical staff, increased use of digital service designs has been recommended by most governments in Scandinavian and European countries. Virtually supported Hospital-at-Home (HaH) models, delivering acute hospital services in-home have been shown to be both feasible and beneficial. Nevertheless, implementation and scaling barriers are major challenges. To enhance implementation of HaH in Scandinavia, the Nordic Digital Health & Education (NorDigHE) project has developed a compre-hensive virtual education on HaH for clinical staff. The present study aims to evaluate the implementation impact of the NorDigHE education embedded in the WHO Fast-track Implementation Model (WHO Fast-IM).

Methods and analysis: We use a randomized design and nested qualitative studies to meet the aim. Via open-call, hospitals will be recruited in Denmark, Norway, and Sweden and randomized to either receive the education embedded in the WHO Fast-IM or to continue treatment as usual. The primary outcome of the RCT is HaH implementation measured at organization level, understood as a change in clinical practice by increased HaH activity. Secondary outcomes are HaH knowledge and motivation among clinical staff as well as patient days in hospital, days hospitalized at home, 30-day readmission, and mortality. Data are collected at baseline, after 3, and 6 months. A 12-month maintenance measurement is performed in the intervention group. Post-study, the control group is offered the NorDigHE education as a participant re-tention measure. In addition, the attitudes, experiences, and preferences of HaH among patients, clinical staff, and management are collected via nested semi-structured interviews.

ELIGIBILITY:
Inclusion criteria:

Hospitals with clinical departments treating acutely ill in-patients that have, or are ready to establish, the prerequisites and infrastructure for HaH - regardless of the specific approach, envisioned HaH model, primary sector collaborations, or local sector collaboration agreements and frameworks. Each hospital must have or be ready to establish:

1. a governance structure to organize and oversee HaH-services.
2. an IT-platform capable of managing data from and to HaH patients.
3. a safe communication pathway between HaH-patient and the hospital.
4. clear agreements on types of data to be exchanged between HaH-patient and hospital.
5. agreements on roles, responsibilities, and capacity (incl. possibly primary sector entities).
6. clinical guidelines, standard operating procedures, and action plans to support the HaH work.

Exclusion Criteria:

* Hospitals that do not have or are not ready to secure relevant pre-requisites listed above (a to f).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HaH implementation | From enrollment until 6 months follow-up measurement
  The primary outcome, HaH implementation at the organizational level, is defined as a change in clinical practice, measured by the proportion of eligible patients who receive HaH.

SECONDARY OUTCOMES:
Staff's motivation | From enrollment until 6 months follow-up
  Staff's motivation to work with HaH. Staff HaH motivation is measured by Intrinsic Motivation Inventory (IMI) Scale questionnaires. Participants will be presented with a series of statements and asked to indicate how true each statement is for them on a 7-point scale, where 1 represents 'not true at all' and 7 represents 'very true'.
Staff's knowledge | From enrollment until 6 months follow-up
  Staff members' knowledge on HaH. Staff's knowledge is collected as pre- and post-education questionnaires at baseline and at 6 months follow-up. The knowledge questionnaires have been developed prior to the study and has undergone pilot-validation with healthcare students, clinical staff, and education sector experts as part of the NorDigHE project.
Days hospitalized at home | From enrollment until 6 months follow-up
  Length of stay while hospitalized at home versus in the hospital. Measured using registry data for patients admitted to the department during trial.
30-day readmission | From enrollment until 6 months follow-up
  The percentage of patients that readmit to the hospital within 30 days with the same illness they were previously discharged. Measured using registry data for patients admitted to the department during the trial.
Mortality | From enrollment until 6 months follow-up
  Tthe number of deaths in participating hospitals (and their departments) during the trial (death rate)

CONTACTS AND LOCATIONS:
Overall Officials: Thea K Fischer, Principal Investigator — Forskningsafdelingen, Nordsjællands Hospital
Locations (3):
- Nordsjællands Hospital, Hillerød, Capitol Region of Denmark, Denmark
- University College of Østfold, Fredrikstad, Østfold fylke, Norway
- Sahlgrenska University hospital, Göteborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Foy R, Ivers NM, Grimshaw JM, Wilson PM. What is the role of randomised trials in implementation science? Trials. 2023 Aug 16;24(1):537. doi: 10.1186/s13063-023-07578-5. PMID 37587521
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294
- [Background] Jakobsen AS, Laursen LC, Rydahl-Hansen S, Ostergaard B, Gerds TA, Emme C, Schou L, Phanareth K. Home-based telehealth hospitalization for exacerbation of chronic obstructive pulmonary disease: findings from "the virtual hospital" trial. Telemed J E Health. 2015 May;21(5):364-73. doi: 10.1089/tmj.2014.0098. Epub 2015 Feb 5. PMID 25654366
- [Background] Sandreva T, Larsen MN, Rasmussen MK, Nielsen TL, von Sydow C, Schmidt TA, Fischer TK. Transforming health care: Investigating Influenzer, a novel telemedicine-supported early discharge program for patients with lower respiratory tract infection: A non-randomized feasibility study. J Telemed Telecare. 2025 Sep;31(8):1138-1151. doi: 10.1177/1357633X241254572. Epub 2024 May 23. PMID 38780386
- [Background] Pietersen PI, Bhatnagar R, Rahman NM, Maskell N, Wrightson JM, Annema J, Crombag L, Farr A, Tabin N, Slavicky M, Skaarup SH, Konge L, Laursen CB. Evidence-based training and certification: the ERS thoracic ultrasound training programme. Breathe (Sheff). 2023 Jun;19(2):230053. doi: 10.1183/20734735.0053-2023. Epub 2023 Jul 11. PMID 37492346
- [Background] Vindrola-Padros C, Singh KE, Sidhu MS, Georghiou T, Sherlaw-Johnson C, Tomini SM, Inada-Kim M, Kirkham K, Streetly A, Cohen N, Fulop NJ. Remote home monitoring (virtual wards) for confirmed or suspected COVID-19 patients: a rapid systematic review. EClinicalMedicine. 2021 Jul;37:100965. doi: 10.1016/j.eclinm.2021.100965. Epub 2021 Jun 23. PMID 34179736
- [Background] Levine DM, Ouchi K, Blanchfield B, Diamond K, Licurse A, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: a Pilot Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):729-736. doi: 10.1007/s11606-018-4307-z. Epub 2018 Feb 6. PMID 29411238
- [Background] Leong MQ, Lim CW, Lai YF. Comparison of Hospital-at-Home models: a systematic review of reviews. BMJ Open. 2021 Jan 29;11(1):e043285. doi: 10.1136/bmjopen-2020-043285. PMID 33514582
- [Background] Ankersen DV, Noack S, Munkholm P, Sparrow MP. E-Health and remote management of patients with inflammatory bowel disease: lessons from Denmark in a time of need. Intern Med J. 2021 Aug;51(8):1207-1211. doi: 10.1111/imj.15132. Epub 2021 Aug 3. PMID 34346152
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] J.K. Svane, L. Konge, and H. Tønnesen, "Fast and Well-reported Implementation: Fast-IM and RE-AIM", Clin. Health Promot. - Res. Best Pract. Patients Staff Community, bd. 10., no. 1, p. 10-14, dec. 2020, doi: 10.29102/clinhp.20003.
- [Background] Svane JK, Chiou ST, Groene O, Kalvachova M, Brkic MZ, Fukuba I, Harm T, Farkas J, Ang Y, Andersen MO, Tonnesen H. A WHO-HPH operational program versus usual routines for implementing clinical health promotion: an RCT in health promoting hospitals (HPH). Implement Sci. 2018 Dec 22;13(1):153. doi: 10.1186/s13012-018-0848-0. PMID 30577871
- [Background] Goncalves-Bradley DC, Iliffe S, Doll HA, Broad J, Gladman J, Langhorne P, Richards SH, Shepperd S. Early discharge hospital at home. Cochrane Database Syst Rev. 2017 Jun 26;6(6):CD000356. doi: 10.1002/14651858.CD000356.pub4. PMID 28651296
- [Background] Wallis JA, Shepperd S, Makela P, Han JX, Tripp EM, Gearon E, Disher G, Buchbinder R, O'Connor D. Factors influencing the implementation of early discharge hospital at home and admission avoidance hospital at home: a qualitative evidence synthesis. Cochrane Database Syst Rev. 2024 Mar 5;3(3):CD014765. doi: 10.1002/14651858.CD014765.pub2. PMID 38438114
- [Background] Edgar K, Iliffe S, Doll HA, Clarke MJ, Goncalves-Bradley DC, Wong E, Shepperd S. Admission avoidance hospital at home. Cochrane Database Syst Rev. 2024 Mar 5;3(3):CD007491. doi: 10.1002/14651858.CD007491.pub3. PMID 38438116
- See also: World Health Organization, Global strategy on human resources for health: workforce 2030. Geneva: World Health Organization, 2016. Seen: 6. juni 2024. — https://iris.who.int/handle/10665/250368
- See also: European Commission, "CORDIS programne: Societal Challenges - Health, demographic change and well-being", EU, H2020-EU.3.1., 2014. [Online]. — https://cordis.europa.eu/programme/id/H2020-EU.3.1.
- See also: NOU: Norges offentlige utredninger, "Tid for handling: Personellet i en bærekraftig helse- og omsorgstjeneste", Departementenes sikkerhets- og serviceorganisasjon Teknisk redaksjon, 2023:4, 2023. [Online]. — https://www.regjeringen.no/contentassets/337fef958f2148bebd326f0749a1213d/no/pdfs/nou202320230004000dddpdfs.pdf
- See also: Kommissionen for robusthed i sundhedsvæsenet, "Robusthedskommissionens anbefalinger", sep. 2023. [Online]. — https://www.ism.dk/Media/638336462586551242/Robusthed-Samlet-Rapport-TILG.pdf
- See also: Socialdepartementet SE, "Effektiv och behovsbaserad digital vård", Ds 2023:27, 2023. [Online]. — https://www.regeringen.se/rattsliga-dokument/departementsserien-och-promemorior/2023/09/ds-202327/
- See also: M. Monalto, "Definition: What is Hospital at Home? | WHAHC", WHAHC-community. Seen: 4. februar 2025. [Online]. — https://whahc-community.kenes.com/mod/page/view.php?id=1042
- See also: "NorDigHE.org", Nordighe. Seen: 4. februar 2025. [Online] — https://www.nordighe.org
- See also: "Skillhabit". Set: 3. februar 2025. [Online]. — https://www.skillhabit.com/
- See also: D. L. Kirkpatrick, "The Kirkpatrick Model", Kirkpatrick Partners, LLC. — https://www.kirkpatrickpartners.com/the-kirkpatrick-model/
- See also: Better use of home monitoring. Experience from five departments of cardiology in the Capital Region of Denmark. — https://www.regionh.dk/patientinddragelse/udgivelser/udgivelser/Documents/Bedre%20brug%20af%20hjemmemonitorering.pdf
- See also: "The Hospital moves into the living room during the pandemic". A.G. Poulsen, 2024 — https://ugeskriftet.dk/nyhed/hospitalet-rykker-hjem-i-stuen-under-epidemien
- See also: "WARD Home Pilot - WARD Project" — https://ward247.org/ward-home-ii/
- See also: "Projects - DEFACTUM - Social, sundhed og arbejdsmarked" — https://www.defactum.dk/
- See also: Erfaringer med Fremskudt akutfunktion på kommunale sengepladser i eHospitalet, Region Sjælland — https://www.vive.dk/media/pure/qz55bmrz/24484546